CLINICAL TRIAL: NCT02938650
Title: Assessing the Role of Nitrosomonas Eutropha on Nitrolipids in the Skin
Brief Title: Nitrosomonas Eutropha on Nitrolipids in the Skin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 916019
Record Dates: First submitted 2016-10-17; First posted 2016-10-19 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Inflammation
Keywords: nitrolipid; microbiome; inflammation; cytokine
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Intervention Model Description: 15 healthy controls will participate in the study Another set of healthy controls (n=20) will be recruited so that they participate in blood draws.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nitrosomonas eutropha spray (Other): Subjects will receive nitrosmonas eutropha spray that they will apply twice a day.
  Interventions: Drug: Nitrosomonas eutropha

INTERVENTIONS:
Drug: Nitrosomonas eutropha — Subjects will get nitrosomonas eutropha to apply for one week. There is only one arm to this study. Subjects will apply the medication twice a day for one week.

SUMMARY:
We are looking to see how the addition of nitrosomonas alters the presence of nitrolipids and inflammatory cytokines on the skin.

DETAILED DESCRIPTION:
We are looking to see how the nitrosomonas alters nitrolipids in the skin and the inflammatory cytokines of the skin.

We will be using healthy subjects over the course of 2 weeks.

Subjects will be using a neutral cleanser for one week prior to the study, skin microbiome,facial photography, lipid and cytokine measurements will be taken at baseline. Subjects will then start using nitrosomonas spray twice daily for one week.

There is a portion of the study where the subjects will have skin microbiome, facial photography, lipid measurements, blood pressure measurements and a bloow draw before and after using the nitrosomonas spray for one week.

ELIGIBILITY:
Inclusion Criteria:

* Those aged 18 and over
* Healthy Subjects with clear skin

Exclusion Criteria:

* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners
* Those with acne, eczema, seborrheic dermatitis, rosacea or polycystic ovarian syndrome
* Those who have started new oral medication in the last four weeks
* Those who have used systemic antibiotics in the last month
* Those who have used isotretinoin in the last 6 weeks
* Those who have used topical antibiotics or retinoid in the last two weeks.
* Those who have autoimmune or metabolic diseases
* Those who have changed brands of oral contraceptive within the last four weeks
* Those who have chronic medical disorders
* Those whose with active skin infections
* Concomitant use of nitrates
* Concomitant use of anti-hypertensive agents
* Those with syncopal episodes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-10; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Alteration in microbiome diversity and species | one week
  We will assess the alteration in the skin microbiome over a one week period by assessing the Shannon Diversity Index
Alteration in nitrolipids in the skin | one week
  we will assess the change in nitrolipid profile of sebum collections from the skin after application of the nitrosomonas spray.

SECONDARY OUTCOMES:
Alteration in skin cytokines | one week
  we will assess the change in skin cytokines with the use of a non-invasive skin collection.
Alteration in blood lipids | one week
  we will assess the change in blood lipids by performing a blood draw
Blood pressure readings | one week
  blood pressure readings will be performed throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Raja K Sivamani, MD, Principal Investigator — UC Davis
Locations (1):
- University of California, Davis Dermatology Clinical Trials Unit, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No